CLINICAL TRIAL: NCT01943422
Title: Dose-seeking and Efficacy Study of the Combination of the BRAF Inhibitor Vemurafenib and High-dose Interferon Alfa-2b for Therapy of Advanced Melanoma
Brief Title: Safety and Efficacy Study of Vemurafenib and High-dose Interferon Alfa-2b in Melanoma
Acronym: 12-107
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: John Kirkwood (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, John Kirkwood, Director of Melanoma Program at UPCI, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-107
Record Dates: First submitted 2013-08-27; First posted 2013-09-17 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Melanoma
Keywords: advanced; melanoma; Vemurafenib; High-dose Interferon alfa-2b
MeSH Terms: conditions — Melanoma | interventions — Interferon alpha-2; Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vemurafenib + IFNα-2b (10 MU/m2/d) (Experimental): Vemurafenib + High-dose Interferon alfa-2b (10 MU/m2/d)
  * IFNα-2b will be administered intravenously for 5 consecutive days (Monday through Friday) every week for 4 weeks (induction)
  * Vemurafenib will be dosed continuously at the standard Food and Drug Administration (FDA) approved dose of 960mg twice a day orally without dose interruption except for toxicities attributable to this agent.
  Interventions: Drug: High-dose Interferon alfa-2b; Drug: Vemurafenib
- Vemurafenib + IFNα-2b(15 MU/m2/d) (Experimental): Vemurafenib + High-dose Interferon alfa-2b (15 MU/m2/d)
  * IFNα-2b will be administered intravenously for 5 consecutive days (Monday through Friday) every week for 4 weeks (induction)
  * Vemurafenib will be dosed continuously at the standard Food and Drug Administration (FDA) approved dose of 960mg twice a day orally without dose interruption except for toxicities attributable to this agent.
  Interventions: Drug: High-dose Interferon alfa-2b; Drug: Vemurafenib
- Vemurafenib + IFNα-2b (20 MU/m2/d) (Experimental): Vemurafenib + High-dose Interferon alfa-2b (20 MU/m2/d)
  * IFNα-2b will be administered intravenously for 5 consecutive days (Monday through Friday) every week for 4 weeks (induction)
  * Vemurafenib will be dosed continuously at the standard Food and Drug Administration (FDA) approved dose of 960mg twice a day orally without dose interruption except for toxicities attributable to this agent.
  Interventions: Drug: High-dose Interferon alfa-2b; Drug: Vemurafenib

INTERVENTIONS:
Drug: High-dose Interferon alfa-2b — •Vemurafenib at standard dosing with a 2 week lead-in period to identify potential effects. IFNα-2b following this (week 2 onwards) at standard induction (4 weeks) and maintenance (48 weeks) doses.
  Other Names: IFNα-2b (HDI)
Drug: Vemurafenib — Vemurafenib is a prescription medicine used to treat melanoma, that has spread to other parts of the body or cannot be removed by surgery, and that has a certain type of abnormal "BRAF" gene.
  Other Names: Zelboraf

SUMMARY:
This is a dose-seeking and efficacy study of combined BRAF Inhibitor Vemurafenib and High-dose Interferon alfa-2b for therapy of advanced melanoma.

DETAILED DESCRIPTION:
* Dose-selection and dose-expansion study of combination therapy with high-dose interferon alfa-2b and vemurafenib.
* Vemurafenib at standard dosing with a 2 week lead-in period to exploit potential immunomodulatory effects. Concurrent HDI following this (week 2 onwards) at standard induction (4 weeks) and maintenance (48 weeks) doses.
* Modified Storer's "up and down" dose escalation schema using 3 fixed dose levels for HDI and a fixed sample size that allows efficient identification of recommended phase II dose.
* 36-63 patients will be enrolled depending on toxicity parameters. oIn the dose-selection portion, 3 patients will be enrolled per dose level, starting from the lowest dose level. Enrollment will occur serially allowing for the observation of toxicity during the observation period.

oIterative enrollment of up to 3 subjects per cohort will be continued until a total of 30 evaluable subjects have been enrolled.

oThe dose level at which the RLT rate is the closest to 1/3 will be considered as RP2D.

oDuring the dose-expansion portion of the trial, depending on the number of patients treated at RP2D during the dose-selection portion, additional patients may be enrolled - the accrual target is 36 patients treated at RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a written informed consent.
* 18 years of age.
* Patients must have histologically confirmed recurrent stage III or stage IV melanoma (AJCC 7th edition classification).
* BRAF V600E and V600K mutated
* Cutaneous squamous cell carcinomas (SCC) lesions identified at baseline must be excised. Adequate wound healing is required prior to study entry.
* Patients must have measurable disease as defined by the Response Evaluation Criteria in Solid Tumors v1.1.
* Patients must have adequate hematologic, renal, and liver function:

  * WBC ≥ 3,000/mm3
  * ANC ≥ 1500
  * Hb ≥ 9g/dL (women) or ≥ 11g/dL (men) (supportive transfusions will be allowed during induction and maintenance phases to maintain these levels)
  * Platelets ≥ 100,000/mm3 (supportive transfusions will be allowed during induction and maintenance phases to maintain these levels)
  * Serum Creatinine ≤ 1.5 x upper limit of normal (ULN)
  * Serum Bilirubin ≤ 1.5 x ULN
  * Serum AST/ALT ≤ 2.5 x ULN
* EKG documenting normal intervals.
* Fully recovered from any effects of major surgery, and be free of significant detectable infection.
* ECOG performance status of 0 or 1.
* Free of active brain metastases by contrast-enhanced CT/MRI scans within 4 weeks prior to starting the study drugs.
* Female patients of child bearing potential must have a negative pregnancy test (within 7 days from the time of randomization).

Exclusion Criteria:

* Serious illnesses, such as: cardiovascular disease (uncontrolled congestive heart failure, uncontrolled hypertension, cardiac ischemia, myocardial infarction, and severe cardiac arrhythmia), bleeding disorders, symptomatic autoimmune diseases, severe obstructive or restrictive pulmonary diseases, uncontrolled endocrine disorders (hypothyroidism, hyperthyroidism and diabetes mellitus), retinopathy, active systemic infections, and inflammatory bowel disorders. This includes known HIV or AIDS-related illness, or active HBV and HCV.
* Prior therapy (except for adjuvant immunotherapy) with a BRAF and/or MEK and/or ERK inhibitors.
* Refractory nausea, vomiting, small bowel resection or any other gastrointestinal ailment that would preclude study drug absorption.
* Cardiac abnormalities

  * Mean QTc interval ≥ 480 msec at screening.
  * Recent ACS/AMI - defined as within 24 weeks prior to screening.
  * Recent PCI/PTCA - defined as within 24 weeks prior to screening.
  * Recent malignant cardiac arrhythmias - all except sinus arrhythmia within 24 weeks prior to screening.
  * Symptomatic heart failure - NYHA Class ≥ II symptoms.
* Active infection or antibiotics within one-week prior to study, including unexplained fever Any significant psychiatric disease, medical intervention, or other condition, which in the opinion of the principal investigator, could prevent adequate informed consent or compromise participation in the clinical trial.
* Systemic steroid or other immunosuppressive therapy within 4 weeks of starting the study.
* Lactating females or pregnant females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events to determine Ph II dose | 12-24 months from study start
  At each dose level, the number of patients experiencing Adverse Events over their course of treatment will be characterized by type of Adverse Event and grade using NCI CTCAE (v4.0), and by time of onset in relation to the first day of therapy.

SECONDARY OUTCOMES:
Progression Free and overall survival (Efficacy) | 48 months
  •Progression Free Survival will be evaluated at 6 months using the Kaplan-Meier method. Overall Survival will be measured from the initial date of treatment to the recorded date of death, and analyzed similarly to Progression Free Survival. Overall Survival will also be analyzed with the Kaplan-Meier method. The complete response rate and partial response rate will be estimated by the proportion of patients with a best response respectively by RECIST criteria.

OTHER OUTCOMES:
Improve tumor STAT signaling | 48 months
  Melanoma metastases removed from patients pretreatment, post-BRAFI alone and Post B-RAF+ will be analyzed for expression of IFNAR1 and immunologically relevant molecules such as HLA antigens, APM components and MA; these results will be correlated with T cell infiltration. In addition the metastases will be tested for extent of melanoma cell proliferation and apoptosis.

CONTACTS AND LOCATIONS:
Overall Officials: John Kirkwood, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States